CLINICAL TRIAL: NCT05388747
Title: Population Pharmacokinetics, Effectiveness and Safety of Cefuroxime in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Tianjin Central Hospital of Gynecology Obstetrics (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2022-PPK-002
Record Dates: First submitted 2022-05-22; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — Cefuroxime

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cefuroxime — Population pharmacokinetics, effectiveness, and safety of cefuroxime

SUMMARY:
Cefuroxime is a time-dependent antibiotic that is used to treat bacterial infections. However, population pharmacokinetic，effectiveness and safety data for cefuroxime in neonates are lacking. The aim of this study was to assess the population pharmacokinetics, effectiveness, and safety of cefuroxime in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Age: postnatal age ≤28 days;
* Cefuroxime used as part of antimicrobial treatment;
* Parental written consent.

Exclusion Criteria:

* Expected survival time less than the treatment cycle;
* Receiving other systemic trial drug therapy;
* Other factors that the researcher considers unsuitable for inclusion.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonatal patients with infections
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-16 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The peak plasma drug concentration of cefuroxime | at (5-10) minutes after intravenous administration
  To detect the peak plasma drug concentration of cefuroxime after intravenous administration.
The random plasma drug concentration of cefuroxime | at (0.25-10) hours after intravenous administration.
  To detect the random plasma drug concentration of cefuroxime after intravenous administration.
The trough plasma drug concentration of cefuroxime | at 1-2 hours before the next administration
  To detect the trough plasma drug concentration of cefuroxime after intravenous administration.
The time of free drug concentration exceeding the minimal inhibitory concentration (fT>MIC) | Through study completion, an average of 3 days
  PD target
Adverse events | Through study completion, an average of 15 days
  Drug-related adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality, China